CLINICAL TRIAL: NCT05341609
Title: A Multicenter, Single-blind, Randomized, Controlled Study to Evaluate the Efficacy and Safety of JT001 (VV116) Compared With Paxlovid for the Early Treatment of COVID-19 in Participants With Mild to Moderate COVID-19
Brief Title: Efficacy and Safety of JT001 (VV116) Compared With Paxlovid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JT001-010-COVID-19
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: JT001(VV116); Mild to Moderate COVID-19
MeSH Terms: conditions — COVID-19 | interventions — GS-621763; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JT001(VV116) (Experimental): Day 1: 600mg, Q12H X 1 day; Day 2~5: 300mg, Q12H X 4 days
  Interventions: Drug: JT001
- Paxlovid (Active Comparator): Day 1~5: 300 mg of Nirmatrelvir and 100 mg of ritonavir, Q12H X 5 days
  Interventions: Drug: Paxlovid

INTERVENTIONS:
Drug: JT001 — Day 1: 600mg, Q12H X 1 day; Day 2~5: 300mg, Q12H X 4 days
  Other Names: VV116
  Arms: JT001(VV116)
Drug: Paxlovid — Day 1~5: 300 mg of Nirmatrelvir and 100 mg of ritonavir, Q12H X 5 days
  Other Names: Nirmatrelvir / ritonavir
  Arms: Paxlovid

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JT001 (VV116) Compared With Paxlovid for the Treatment of Coronavirus Disease 2019 (COVID-19) in Participants With Mild to Moderate COVID-19.

DETAILED DESCRIPTION:
Screening Interested participants will sign the appropriate informed consent form (ICF) prior to completion of any study procedures.

The investigator will review symptoms, risk factors and other non-invasive inclusion and exclusion criteria prior to any invasive procedures.

Treatment and Assessment Period

This is the general sequence of events during the 28-day treatment and assessment period:

Complete baseline procedures Participants are randomized to an intervention group Participants receive study intervention (Q12H X 5 days), and Complete all safety monitoring

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a positive SARS-CoV-2 test result.
* Participants who have one or more mild or moderate COVID-19 symptoms, and total symptom score ≥ 2.
* Participants who have one or more of the following requirements: ≤7 days from the first positive test for SARS-COV-2 virus infection to the first dose; ≤5 days from the first onset of COVID-19 symptoms to the first dose; SARS-CoV-2 Ct Value ≤20 within 24 hours prior to the first dose.
* Participants who satisfy one or more than one of the following high risks for progression to severe COVID-19, including death.
* Participants who must agree to adhere to contraception restrictions.
* Participants who understand and agree to comply with planned study procedures.
* Participants or legally authorized representatives can give written informed consent approved by the Ethical Review Board governing the site.
* Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participants who are judged by the investigator as likely to progress to severe/critical COVID-19 prior to randomization.
* Participants who have SpO2≤93% on room air at sea level or PaO2/FiO2≤ 300, or respiratory rate ≥30 per minute.
* Participants who require mechanical ventilation or anticipated impending need for mechanical ventilation.
* Participants who have eye disease.
* Participants who have any of the following conditions when screening: ALT or AST>1.5 ULN; e GFR <60 mL/min.
* Participants who have known allergies to any of the components used in the formulation of the interventions.
* Any medical condition, which in the opinion of the Investigator, will compromise the safety of the participant.
* Participants who have received a SARS-CoV-2 monoclonal antibody treatment or prevention, or antiviral treatment (including the investigational treatment).
* Participants who have received convalescent COVID-19 plasma treatment.
* Participant's use of contraindicated drugs in the Package Insert of Nirmatrelvir Tablet/Ritonavir Tablets.
* Participants who have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed.
* Participants who are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Female who is pregnant or breast-feeding or plan to be pregnant within this study period.
* Male whose wife or partner plan to be pregnant within this study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Time to sustained clinical recovery | Up to 28 days
  Time to sustained clinical recovery up to 28 days.

SECONDARY OUTCOMES:
AEs and SAEs through Day 28 | Up to 28 days
  AEs and SAEs through Day 28
Percentage of participants who experience these events by Day 28 | Day 1 to 28 days
  Percentage of participants who experience these events by Day 28
  Progress to severe and/or critical COVID-19; Death from any cause
Percentage of clinical recovery participants | Days 3, 5, 7, 10, 14, 21 and 28
  Percentage of clinical recovery participants from baseline to Days 3, 5, 7, 10, 14, 21 and 28
The change of COVID-19 symptom scores | Days 3, 5, 7, 10, 14, 21 and 28
  The change of "COVID-19 symptom scores" from baseline to Days 3, 5, 7, 10, 14, 21 and 28, the score ranges from 0 to 33 and higher scores mean a worse symptom.
The change of WHO clinical progression scale | Days 3, 5, 7, 10, 14, 21 and 28
  The change of "WHO clinical progression scale" from baseline to Days 3, 5, 7, 10, 14, 21 and 28, the score ranges from 0 to 10 and higher scores mean a worse clinical progression.
Percentage of participants with SARS-CoV-2 clearance | Days 3, 5, 7, 10, 14
  Percentage of participants with SARS-CoV-2 clearance on Days 3, 5, 7, 10 and 14
The change of SARS-COV-2 Ct value | Days 3, 5, 7, 10, 14
  The change of SARS-COV-2 Ct value at Days 3, 5, 7, 10, 14
The change of Chest CT scan | Days 7 or 10
  The change of Chest CT scan from baseline to Days 7 or 10. The change from baseline involves not changed, getting worse, getting better as assessed by the investigator.
Percentage of the participants who have progression of COVID-19 though Day 28 | Up to 28 days
  Progress to severe and/or critical COVID-19; Death from any cause
Percentage of participants whose "WHO clinical progression scale" reduced at least one level | Days 3, 5, 7, 10, 14, 21 and 28
  Percentage of participants whose "WHO clinical progression scale" reduced at least one level from baseline to Days 3, 5, 7, 10, 14, 21 and 28. The score ranges from 0 to 10 and the higher scores mean a worse clinical progression level.
Time to sustained clinical symptom resolution | Up to 28 days
  Time to sustained clinical symptom resolution
Percentage of participants with clinical symptom resolution | Days 3, 5, 7, 10, 14, 21 and 28
  Percentage of participants with clinical symptom resolution from baseline to Days 3, 5, 7, 10, 14, 21 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (7):
- China (7):
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - ShuGuang Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Z, Gao W, Bao H, Feng H, Mei S, Chen P, Gao Y, Cui Z, Zhang Q, Meng X, Gui H, Wang W, Jiang Y, Song Z, Shi Y, Sun J, Zhang Y, Xie Q, Xu Y, Ning G, Gao Y, Zhao R. VV116 versus Nirmatrelvir-Ritonavir for Oral Treatment of Covid-19. N Engl J Med. 2023 Feb 2;388(5):406-417. doi: 10.1056/NEJMoa2208822. Epub 2022 Dec 28. PMID 36577095